CLINICAL TRIAL: NCT02168244
Title: Reduction of Injection-related Pain Caused by Subcutaneous Administration of Biologic Drugs in Psoriasis
Brief Title: Reduction of Pain Caused by Biologic Drugs in Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 14-0535
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Psoriasis; Pain
Keywords: psoriasis; biologics; subcutaneous; pain; heat; ice
MeSH Terms: conditions — Psoriasis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ice pack (Active Comparator): Pre-treatment with ice - Ice applied to the skin 2-3 minutes before injecting biologic drug injection
  Interventions: Other: Ice pack
- Heating Pack (Active Comparator): Pre-treatment with heat - Heat applied to the skin 2-3 minutes before injecting biologic drug injection
  Interventions: Other: Heating Pack
- No treatment before injection (No Intervention): No treatment applied to the skin 2-3 minutes before injecting biologic drug injection

INTERVENTIONS:
Other: Heating Pack — Application of heat to skin for 2-3 minutes prior to injection of biologic drug
  Arms: Heating Pack
Other: Ice pack — Application of cold to skin for 2-3 minutes prior to injection of biologic drug
  Arms: Ice pack

SUMMARY:
Injectable biologic drugs are used as a treatment of psoriasis. These injections can sometimes be associated with pain. In this study the investigators aim to reduce the pain by applying heat or ice to the skin 2-3 minutes before injecting the drug, and to compare the pain to injection without any heat or ice.

DETAILED DESCRIPTION:
As part of their therapy, some patients with psoriasis require treatment with biologic drugs, which are injected into their skin. While these are very effective, patients may experience some pain or discomfort associated with the injection of these drugs.

In this research study conducted at Mount Sinai hospital, the investigators aim to identify whether this injection-related pain can be reduced if the area of skin to be injected with the biologic drug is treated with either ice packs or heating for two to three minutes prior to the injection.

The investigators' aim is to include a total of 110 patients into this study, who have been started by their physician on one of these biologic drugs, such as etanercept, adalimumab, ustekinumab, or receiving secukinumab as part of a research study. Patients will be recruited at the Dermatology department. Patients who are receiving a biologic drug, which is injected subcutaneously (into their skin) are eligible to participate in this study.

Each patient will receive his/her injection at our study site, by a study doctor/investigator. The same designee should inject the subject all three times. Each patient will receive a total of three of their biologic drug injections at the study site, so he/she can receive the injection once following pre-treatment with ice, once following pre-treatment with heating, and once without any pre-treatment.

Patients will then be asked to mark the intensity of the pain associated with the injection on a scale, consisting of a horizontal line, by placing a single mark on the scale. The order of pre-treatment with ice or heat, or no pre-treatment will be randomized among all subjects (1/3 will receive ice first, 1/3 will receive heat first, 1/3 will receive no treatment first; the same randomization ratio will apply for the second and third injections).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring treatment with a biologic drug
* Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give written, signed and dated informed consent before any study-related activity is performed

Exclusion Criteria:

* Patients receiving concurrent therapeutic injections for other indications
* Patients who have taken analgesics within 12 hours of their injection
* A past history of cold-, heat- or pressure-induced urticaria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduction of pain measured on a visual analogue scale | At time of injection

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States